CLINICAL TRIAL: NCT05800899
Title: Stage II Efficacy Trial of a Culturally Informed Brief Intervention to Reduce Alcohol Related Health Disparities and Treatment Inequities Among Latinxs
Brief Title: Trial of a Culturally Informed Brief Intervention to Reduce Alcohol Related Health Disparities and Treatment Inequities Among Latinxs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Collaborators: University of Texas at Austin (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); El Paso County General Hospital dba University Medical Center (Unknown)
Responsible Party: Principal Investigator, Craig Field, Principal Investigator, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTexasElPaso
Record Dates: First submitted 2023-02-23; First posted 2023-04-06 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use Disorder
Keywords: Brief Motivational Intervention; Cultural Adaptation; Mechanisms of Change; Self-Determination Theory; Harm Reduction; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism; Harm Reduction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Research staff conducting the initial assessment prior to randomizations to brief interventions or culturally informed intervention and those conducting follow-up assessments will be blind to participant assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Motivational Interviewing (Active Comparator)
  Interventions: Behavioral: Brief Motivational Interviewing
- Culturally Adaptation Brief Motivational Interviewing (Experimental)
  Interventions: Behavioral: Culturally adaptation brief motivational interviewing

INTERVENTIONS:
Behavioral: Brief Motivational Interviewing — Standard non-adapted brief motivational interviewing based on motivational interviewing.
  Arms: Brief Motivational Interviewing
Behavioral: Culturally adaptation brief motivational interviewing — culturally adapted brief motivational interviewing based on motivational interviewing.
  Arms: Culturally Adaptation Brief Motivational Interviewing

SUMMARY:
This Stage II Randomized Efficacy Trial will compare the effectiveness of a theoretically informed and culturally responsive brief motivational intervention to a non-adapted brief intervention among non-treatment seeking Latinxs admitted for medical treatment of an injury who engage in at risk drinking or were drinking at the time of their injury. The culturally informed brief motivational intervention (CI-BMI) increases autonomous motivation to engage in protective drinking behavior and reduce alcohol problems while addressing barriers to help seeking and facilitating treatment utilization. This project will address the alcohol related health disparities and treatment inequities among Latinx who are more likely to experience alcohol problems yet less likely to receive treatment in order to reduce the negative public health impact of alcohol.

DETAILED DESCRIPTION:
Our prior Stage III Randomized Clinical Trial (n=1496) evaluating ethnic differences in response to brief intervention showed that, compared to non-Latinxs Whites, Latinxs were more likely to reduce alcohol use in response to standard brief alcohol interventions that are not adapted to be culturally responsive (NA-BMI) versus treatment as usual1. In Stage I Community Based Participatory Research (Stage I CBPR), we developed a culturally informed brief motivational intervention (CI-BMI) which adopts a harm reduction approach and focuses on reducing alcohol problems and increasing treatment utilization 2. Through a flexible core approach, CI-BMI introduces substantial modifications to standard brief alcohol interventions to be culturally responsive and is theoretically grounded in self-determination theory (SDT)3-5. The result of Stage I CBPR was CI-BMI which 1) leverages cultural values and strengths while addressing the process of acculturation and acculturative stress; 2) is explicitly designed to meet the basic psychological needs of autonomy, relatedness, and competence by supporting autonomy to enhance autonomous motivation to change drinking behavior; and 3) focuses on harm reduction. Our Stage I CBPR (n=87) demonstrated that CIBMI is feasible and acceptable in pretesting in a Level I Trauma Center5. We hypothesize that CI-BMI will lead to increased engagement in protective drinking behaviors, fewer alcohol problems as well as reduce barriers to help seeking and increase treatment utilization among underserved, non-treatment seeking Latinxs who engage in at risk drinking and are seriously injured. The proposed Stage II Efficacy Trial of CI-BMI will randomize 600 Latinxs admitted to a Level I Trauma Center at University Medical Center in El Paso, Texas to either NA-BMI or CI-BMI conducted by research staff from The University of Texas El Paso. Following admission for medical treatment of an injury, eligible Latinx patients will be those who screen positive for drinking at the time of their injury or engage in at risk drinking. The primary aims of the proposed study are to

1) test the efficacy of CI-BMI in comparison to NA-BMI on alcohol related harm reduction behaviors, alcohol problems, barriers to help seeking and treatment utilization among non-treatment seeking Latinxs and 2) examine the theoretically informed mechanism of behavior change based on SDT including providing autonomy support to meet the basic psychological needs that enhance autonomous motivation. Because the psychological processes underlying the intrasession mechanisms of change remain poorly understood, CI-BMI based on SDT will significantly advance the science and practice of brief interventions6. In addition, planned secondary data analysis will assess the influence of multi-dimensional acculturation/enculturation orientations and acculturative stress on alcohol related outcomes. The results of this study will lead to a theoretically informed and culturally response brief motivation intervention with enhanced generalizability to effectively address alcohol related health disparities and treatment inequities among non-treatment seeking Latinxs.

ELIGIBILITY:
Inclusion Criteria:

* Admission to a level 1 -trauma center
* Involved in a alcohol-related injury
* Self-identify as Latinx
* 18 or older
* Minimum Blood Alcohol Concentration (BAC) score of .001 and/or at risk drinking

Exclusion Criteria:

* Traumatic brain injury or otherwise debilitating injury as indicated by a Glasgow Coma Scale score of less than 15.
* Cognitive impairment as indicated by a score of 24 or less on the Mini-Mental Status Exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in protective drinking strategies on 7-point Protective Behavioral Strategies Scale (PBSS) at 3-month | Baseline and 3 month
  The 20-item Protective Behavioral Strategies Scale (PBSS) will be used to quantify the engagement in harm reduction behaviors which will be assessed at baseline, three, six and twelve month follow up. The PBSS consists of three subscales that reflect different types of strategies: stopping/limiting drinking (7 items), manner of drinking (5 items), and serious harm reduction (3 items). Participants are instructed to rate the degree to which they engage in PBS on a 6-point response scale ranging from 1 (Never) to 6 (Always). change=(3 month -baseline score)
Change from baseline in protective drinking strategies on 7-point Protective Behavioral Strategies Scale (PBSS) at 6-month | Baseline and 6 month
  The 20-item Protective Behavioral Strategies Scale (PBSS) will be used to quantify the engagement in harm reduction behaviors which will be assessed at baseline, three, six and twelve month follow up. The PBSS consists of three subscales that reflect different types of strategies: stopping/limiting drinking (7 items), manner of drinking (5 items), and serious harm reduction (3 items). Participants are instructed to rate the degree to which they engage in PBS on a 6-point response scale ranging from 1 (Never) to 6 (Always). change=(6 month -baseline score)
Change from baseline in protective drinking strategies on 7-point Protective Behavioral Strategies Scale (PBSS) at 12-month | Baseline and 12 month
  The 20-item Protective Behavioral Strategies Scale (PBSS) will be used to quantify the engagement in harm reduction behaviors which will be assessed at baseline, three, six and twelve month follow up. The PBSS consists of three subscales that reflect different types of strategies: stopping/limiting drinking (7 items), manner of drinking (5 items), and serious harm reduction (3 items). Participants are instructed to rate the degree to which they engage in PBS on a 6-point response scale ranging from 1 (Never) to 6 (Always). change=(12 month -baseline score)
change from baseline in alcohol problems on a 5-point scale using the Short Index of Problems (SIP) at 3 months | Baseline and 3 month
  Participants are asked to indicate how often they have experienced each of 15 consequences listed in the items. Each item is responded to on a 5-point response scale ranging from 0 (Never) to 4 (Daily or almost daily). The 15 items will be summed to create a total score. Change = (3-month -baseline score)
change from baseline in alcohol problems on a 5-point scale using the Short Index of Problems (SIP) at 6 months | Baseline and 6 month
  Participants are asked to indicate how often they have experienced each of 15 consequences listed in the items. Each item is responded to on a 5-point response scale ranging from 0 (Never) to 4 (Daily or almost daily). The 15 items will be summed to create a total score. Change = (6 -month -baseline score)
change from baseline in alcohol problems on a 5-point scale using the Short Index of Problems (SIP) at 12 months | Baseline and 12-month
  Participants are asked to indicate how often they have experienced each of 15 consequences listed in the items. Each item is responded to on a 5-point response scale ranging from 0 (Never) to 4 (Daily or almost daily). The 15 items will be summed to create a total score. Change = (12-month -baseline score)

SECONDARY OUTCOMES:
Change from baseline in Attitudes Towards alcohol Treatment Services using the Barriers to Help Seeking Scale (BSAT) at 3 months | Baseline and 3-month
  To asses an individuals attitudes towards alcohol services and treatment the Barriers to Help Seeking Scale (BSAT) measure will be used. The measure utilizes 53 total questions and consist of ten different domains (alcohol treatment, drinking goals, cultural background, immigration, drinking perceptions, feelings towards alcohol treatment services, friends and family, accessing services, life responsibilities, and treatment seeking). Each subscale is summed for a total subscale score (1 strongly agree to 5 strongly disagree). Change = (3month -baseline score)
Change from baseline in Attitudes Towards alcohol Treatment Services using the Barriers to Help Seeking Scale (BSAT) at 6 months | Baseline and 6-month
  To asses an individuals attitudes towards alcohol services and treatment the Barriers to Help Seeking Scale (BSAT) measure will be used. The measure utilizes 53 total questions and consist of ten different domains (alcohol treatment, drinking goals, cultural background, immigration, drinking perceptions, feelings towards alcohol treatment services, friends and family, accessing services, life responsibilities, and treatment seeking). Each subscale is summed for a total subscale score (1 strongly agree to 5 strongly disagree). Change = (6 month -baseline score)
Change from baseline in Attitudes Towards alcohol Treatment Services using the Barriers to Help Seeking Scale (BSAT) at 12 months | Baseline and 12-month
  To asses an individuals attitudes towards alcohol services and treatment the Barriers to Help Seeking Scale (BSAT) measure will be used. The measure utilizes 53 total questions and consist of ten different domains (alcohol treatment, drinking goals, cultural background, immigration, drinking perceptions, feelings towards alcohol treatment services, friends and family, accessing services, life responsibilities, and treatment seeking). Each subscale is summed for a total subscale score (1 strongly agree to 5 strongly disagree). Change = (12 month -baseline score)
change from baseline in treatment utilization using the National Epidemiological Study of Alcohol and Related Conditions (NESARC-III) at 3 months | Baseline and 3-month
  Participants are first asked, "Have you ever gone anywhere or seen anyone for a reason that was related in any way to your drinking - a physician, counselor, Alcoholics Anonymous, or any other community agency or professional?" Participants who respond yes to this first item are told, "I am going to read you a list of community agencies and professionals. For each one, please tell me if you have ever gone for any reason related to your drinking." A list of thirteen types of treatment providers are listed. The 13 items will be summed to create a total score. Change = (3month -baseline score)
change from baseline in treatment utilization using the National Epidemiological Study of Alcohol and Related Conditions (NESARC-III) at 6 months | Baseline and 6-month
  Participants are first asked, "Have you ever gone anywhere or seen anyone for a reason that was related in any way to your drinking - a physician, counselor, Alcoholics Anonymous, or any other community agency or professional?" Participants who respond yes to this first item are told, "I am going to read you a list of community agencies and professionals. For each one, please tell me if you have ever gone for any reason related to your drinking." A list of thirteen types of treatment providers are listed. The 13 items will be summed to create a total score. Change = (6 month -baseline score)
change from baseline in treatment utilization using the National Epidemiological Study of Alcohol and Related Conditions (NESARC-III) at 12 months | Baseline and 12-month
  Participants are first asked, "Have you ever gone anywhere or seen anyone for a reason that was related in any way to your drinking - a physician, counselor, Alcoholics Anonymous, or any other community agency or professional?" Participants who respond yes to this first item are told, "I am going to read you a list of community agencies and professionals. For each one, please tell me if you have ever gone for any reason related to your drinking." A list of thirteen types of treatment providers are listed. The 13 items will be summed to create a total score. Change = (12 month -baseline score)

OTHER OUTCOMES:
Change from baseline in quality of life using the World Health Organization Quality of Life (WHOQoL) at 6 months | Baseline and 6-month
  Quality of life will be assessed using the World Health Organization Quality of Life (WHOQoL) using This allows us to measure to assess quality of life (QOL) within the context of an individual's culture, values system, personal goals, standards and concerns. The measure has 26 items (1 never to 5 always). Items are summed for a total score. Change = (6 month -baseline score)
change from baseline in Basic psychological needs will be assessed using Basic Psychological Need Satisfaction and Frustration Scale (BPNSNF) at 3 months | Baseline and 3-month
  The BPNSNF assesses the satisfaction and frustrations of basic psychological needs as defined by Self Determination Theory including autonomy, competence and relatedness. A total of 24 items are used to assess the satisfaction and frustration of each of the three basic psychological needs. Participants are asked to indicate the degree to which a statement about different kinds of experiences in their life. Participants respond on a five-point Likert scale ranging from not true at all to completely true. A total score is created by subtracting the total score from the three frustration subscales (one for each basic psychological need) from the total score of the three satisfaction subscales (one for each basic psychological need) to get an overall score of basic psychological needs. Change = (3month -baseline score)
change from baseline in Basic psychological needs will be assessed using Basic Psychological Need Satisfaction and Frustration Scale (BPNSNF) at 3 months | Baseline and 6-month
  The BPNSNF assesses the satisfaction and frustrations of basic psychological needs as defined by Self Determination Theory including autonomy, competence and relatedness. A total of 24 items are used to assess the satisfaction and frustration of each of the three basic psychological needs. Participants are asked to indicate the degree to which a statement about different kinds of experiences in their life. Participants respond on a five-point Likert scale ranging from not true at all to completely true. A total score is created by subtracting the total score from the three frustration subscales (one for each basic psychological need) from the total score of the three satisfaction subscales (one for each basic psychological need) to get an overall score of basic psychological needs. Change = (6 month -baseline score)
change from baseline in Basic psychological needs will be assessed using Basic Psychological Need Satisfaction and Frustration Scale (BPNSNF) at 12 months | Baseline and 12-month
  The BPNSNF assesses the satisfaction and frustrations of basic psychological needs as defined by Self Determination Theory including autonomy, competence and relatedness. A total of 24 items are used to assess the satisfaction and frustration of each of the three basic psychological needs. Participants are asked to indicate the degree to which a statement about different kinds of experiences in their life. Participants respond on a five-point Likert scale ranging from not true at all to completely true. A total score is created by subtracting the total score from the three frustration subscales (one for each basic psychological need) from the total score of the three satisfaction subscales (one for each basic psychological need) to get an overall score of basic psychological needs. Change = (12 month -baseline score)
Changes in drinking from baseline using the Drinking Behavior Regulatory Style Questionnaire at 3 month. | Baseline and 3-month
  The measure was designed around Self-determination theories motivational regulations regarding stages of change (amotivation, external regulation, introjected regulation, identified regulation, and integrated regulation). The measure has a total of 53 items and consist of a 7 point-Likert scale ranging from 0 (not true at all) to 7 (very true). Change = (3 month -baseline score)
Changes in drinking from baseline using the Drinking Behavior Regulatory Style Questionnaire at 6 month. | Baseline and 6-month
  The measure was designed around Self-determination theories motivational regulations regarding stages of change (amotivation, external regulation, introjected regulation, identified regulation, and integrated regulation). The measure has a total of 53 items and consist of a 7 point-Likert scale ranging from 0 (not true at all) to 7 (very true). Change = (6 month -baseline score)
Changes in drinking from baseline using the Drinking Behavior Regulatory Style Questionnaire at 12 month. | Baseline and 12-month
  The measure was designed around Self-determination theories motivational regulations regarding stages of change (amotivation, external regulation, introjected regulation, identified regulation, and integrated regulation). The measure has a total of 53 items and consist of a 7 point-Likert scale ranging from 0 (not true at all) to 7 (very true). Change = (12 month -baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: Deidra Roach, PhD, Study Chair — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- University Medical Center of El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
NIAAA Data Archive (NIAAADA)
  Per NOT-AA-22-003, the National Institute on Alcohol Abuse and Alcoholism (NIAAA) expects investigators with applicable grant applications to include plans for sharing NIAAA-funded human subjects grant-related data with the NIAAA Data Archive (NIAAADA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: NIAAA automatically makes study information and data available two years after the study completion date.
Access Criteria: In order to access NIAAA data sharing, users must be an authorized Researcher Auth Service (RAS)
URL: https://nda.nih.gov/niaaa/